CLINICAL TRIAL: NCT06068842
Title: International Real-World Study of MET Overexpression in Patients With Non-Small Cell Lung Cancer
Brief Title: A Study to Assess Prevalence of a Specific Protein Overexpression in Adult Participants With Non-Small Cell Lung Cancer
Acronym: METRIX
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H24-281
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Telisotuzumab Vedotin; ABBV-399; Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Undergoing Chart Review: Participants treated for non small cell lung cancer undergoing chart review and retrospective mesenchymal epithelial transition (MET) overexpression (OE) testing of tissue biopsies.

SUMMARY:
Non-small cell lung cancer (NSCLC) is the most common type of lung cancer, accounting for 80%-85% of lung cancers cases of which 60% are non-squamous (NSQ). This study will evaluate the prevalence of mesenchymal epithelial transition (MET) overexpression (OE) in adult participants with advanced or metastatic NSQ NSCLC.

Archived tissue biopsies will be tested for MET OE and data from approximately 500 participants will be collected. No participants will be enrolled in this study.

Participants' charts will be reviewed. No drug will be administered as a part of this study. The duration of the study will be approximately 15 months.

There is no additional burden for participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Previously consented and/or prospective collection of consent for research use of banked biological materials and clinical data.
* Confirmed advanced and/or metastatic non-squamous (NSQ) non-small cell lung cancer (NSCLC).
* Has formalin-fixed paraffin-embedded (FFPE) tissue collected since 2019.

Exclusion Criteria:

* Specimens collected before 2019.
* Insufficient specimen tissue for testing.
* Insufficient specimen quality (e.g., not 4-5 µm in thickness) which precludes testing.
* Adenosquamous and sarcomatous histologies of NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with non-small cell lung cancer (NSCLC) advanced or metastatic non-squamous (NSQ) NSCLC with available tissue specimens.
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of Mesenchymal Epithelial Transition (MET) protein overexpression (OE) | Up to 15 Months
  OE is defined as: positive: >= 25% of tumor cells with 3+ staining intensity, or negative: < 25% of tumor cells with 3+ staining intensity. High overexpression (OE high) is defined as: positive: >= 50% of tumor cells with 3+ staining intensity negative: < 50% of tumor cells with 3+ staining intensity. These are determined by an immunohistochemistry (IHC) performed by the local laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (19):
- Argentina (2):
  - Hospital Italiano de Buenos Aires /ID# 256999, Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
  - Instituto Alexander Fleming /ID# 256295, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
- Brazil (2):
  - Irmandade da Santa Casa de Misericordia de Porto Alegre /ID# 256487, Porto Alegre, Rio Grande do Sul
  - Hospital Alemao Oswaldo Cruz /ID# 256486, São Paulo
- Canada (3):
  - Nova Scotia Health Authority /ID# 256950, Halifax, Nova Scotia
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université L /ID# 257872, Québec, Quebec
  - Royal University Hospital /ID# 261272, Saskatoon, Saskatchewan
- West China Hospital, Sichuan University /ID# 256906, Chengdu, Sichuan, China
- Rambam Health Care Campus /ID# 256546, Haifa, H_efa, Israel
- Japan (2):
  - Kindai University Hospital /ID# 257890, Osakasayama-shi, Osaka
  - National Cancer Center Hospital /ID# 257889, Chuo-ku, Tokyo
- The Catholic University of Korea, Yeouido ST. Mary's Hospital /ID# 261511, Seoul, Seoul Teugbyeolsi, South Korea
- UOMi Cancer Center - Clinica Tres Torres /ID# 261212, Barcelona, Spain
- Switzerland (2):
  - Universitätsspital Basel /ID# 256677, Basel Town, Canton of Basel-City
  - University Hospital Zurich /ID# 256678, Zurich, Canton of Zurich
- National Taiwan University Hospital /ID# 261542, Taipei City, Taipei, Taiwan
- Burjeel Medical City /ID# 259407, Abu Dhabi, United Arab Emirates
- United Kingdom (2):
  - Queen's University Belfast /ID# 258458, Belfast, Northern Ireland
  - University Hospitals Birmingham NHS Foundation Trust /ID# 260991, Birmingham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=H24-281